CLINICAL TRIAL: NCT01869387
Title: Improvement of Respiratory Muscle Function With Noninvasive Ventilation in Exacerbated COPD Patients Presenting Hypercapnic Respiratory Failure Without Acidosis
Brief Title: Respiratory Muscle Function in COPD Exacerbations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRISOL-MARTINA-2013
Record Dates: First submitted 2013-05-27; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment (No Intervention): Standard treatment consists in bronchodilator and parenteral corticosteroids and oxygen therapy.
- Standard treatment plus non-invasive ventilation (Experimental): This arm consists in bronchodilator and parenteral corticosteroids and oxygen therapy plus non-invasive ventilation.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation
  Arms: Standard treatment plus non-invasive ventilation

SUMMARY:
There is evidence that noninvasive mechanical ventilation (NIV) is effective in the treatment of severe exacerbations of COPD presenting respiratory acidosis.

The aim of the study is to evaluate the benefit of adding NIV to conventional treatment in patients with COPD exacerbation and hypercapnic respiratory failure without acidosis requiring hospital admission. It is known that NIV improves respiratory mechanics, so the primary outcome will be respiratory muscle function.

All patients admitted to the hospital for COPD exacerbation and hypercapnic respiratory failure without acidosis will be included for a period of 12 months. The patients will be randomized into two groups (conventional treatment or conventional treatment plus NIV). Clinical data, blood gases, muscle strength parameters will be collected at the inclusion time and 24h after starting NIV. Quality of life and hospital stay will be measured at discharge. All patients will be followed for a year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to international guidelines ( GOLD)
* COPD exacerbation requiring hospitalization
* Initial blood gases: PaCO2> 50 mm Hg and pH> 7.35.
* If the patient does not have COPD diagnosis at the time of inclusion, it could be included if the diagnosis is confirmed within three months after the exacerbation.

Exclusion Criteria:

* Patients with a pH below 7.35
* Patients with intubation criteria
* Other chronic respiratory diseases (fibrothorax, cystic fibrosis, significant ribcage alterations)
* Neuromuscular Diseases
* Significant associated chronic systemic diseases (severe liver disease, chronic renal failure requiring dialysis, severe heart disease and active neoplasia)
* COPD exacerbation secondary to pulmonary embolism, pneumonia or pneumothorax
* Patients in active treatment with CPAP or home ventilation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle function. | At baseline, at discharge (average of 8 days), 6 months and one year later.
  Measurement of maximal inspiratory pressure and sniff nasal inspiratory pressure using a portable respiratory pressure meter.

SECONDARY OUTCOMES:
Days of hospitalization. | At discharge (average of 8 days).
Dyspnea scale questionnaire | At baseline, at discharge, 6 months and one year later.
Quality of life | At baseline, 6 months and one year later.
Blood gases | At baseline and at discharge (average of 8 days).
Number of hospital readmissions in the next year | At one year after discharge (average of 8 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar (Servei de Pneumología), Barcelona, Barcelona, Spain